CLINICAL TRIAL: NCT04418895
Title: Biomarkers and Clinical Outcomes in Localized Rectal Adenocarcinoma Treated With Neoadjuvant Therapy
Brief Title: Neoadjuvant Therapy for Localized Rectal Adenocarcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of resources
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1933
Record Dates: First submitted 2020-06-02; First posted 2020-06-05 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Rectal Adenocarcinoma
MeSH Terms: conditions — Rectal Neoplasms | interventions — Chemoradiotherapy; Leucovorin; Fluorouracil; Oxaliplatin; XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm: Standard of Care (Experimental): Investigator's choice of total neoadjuvant therapy (TNT) comprised of neoadjuvant chemotherapy and chemoradiation followed by surgical resection; or neoadjuvant chemoradiation followed by surgical resection and then adjuvant chemotherapy.
  Interventions: Other: Chemoradiation; Radiation: short course radiation therapy; Drug: mFOLFOX6; Drug: CAPOX; Drug: fluoropyrimidine +/- oxaliplatin

INTERVENTIONS:
Other: Chemoradiation — Subjects will receive neoadjuvant chemoradiation per standard of care. This is typically comprised of radiotherapy of 5040 cGy (centigray) with concurrent capecitabine 825 mg/m2 by mouth (po) two times daily (bid) (typically rounded to the nearest 500 mg dose) or infusional 5-fluorouracil (5FU). However, dosing and administration are at the discretion of the treating medical and radiation oncologist.
Radiation: short course radiation therapy — An acceptable alternative approach is short-course radiation therapy per standard of care, which is typically comprised of radiotherapy of 25 Gy (gray) in 5 fractions, with surgery within 1 week of completion of therapy or delayed for 6-8 weeks. Selection of the optimal radiation therapy approach is at the discretion of the treating medical oncologist, radiation oncologist, and surgical oncologist. However, generally, short-course radiation therapy is not recommended for low-lying tumors less than 5 centimeters (cm) from the anal verge.
Drug: mFOLFOX6 — possible consolidative neo-adjuvant chemotherapy. This treatment is at the discretion of the treating medical oncologist, radiation oncologist, and surgical oncologist.
  Other Names: leucovorin calcium (folinic acid), fluorouracil, and oxaliplatin
Drug: CAPOX — possible consolidative neo-adjuvant chemotherapy. This treatment is at the discretion of the treating medical oncologist, radiation oncologist, and surgical oncologist.
  Other Names: Capecitabine, Oxaliplatin
Drug: fluoropyrimidine +/- oxaliplatin — possible adjuvant chemotherapy regimen. Subjects who do not receive preoperative mFOLFOX6 or CAPOX typically receive postoperative adjuvant chemotherapy with a fluoropyrimidine +/- oxaliplatin for an additional 16-18 weeks of therapy, if permitted based on recovery after surgical resection and post-surgical performance status. This treatment is at the discretion of the treating medical oncologist. Subjects will remain on study regardless of postoperative therapy administration or duration.

SUMMARY:
This study is a prospective, single-arm, single-center study of investigator's choice of total neoadjuvant therapy (TNT) or neoadjuvant chemoradiation in locally advanced rectal cancer. The standard of care for rectal adenocarcinomas that are triiodothyronine-thyroxine (T3-T4) or node positive has generally been comprised of neoadjuvant chemoradiation, followed by surgical resection and then adjuvant chemotherapy. More recently, TNT, comprised of neoadjuvant chemotherapy and chemoradiation followed by surgical resection, has been increasingly used as a standard therapy approach. While the use of TNT is increasingly common, prospective study of outcomes following TNT has been limited. Moreover, there are not any biomarkers known at this time that impact clinical decision-making or personalization of therapy in the treatment of rectal cancer. In this study, we will collect pre-treatment rectal adenocarcinoma specimens and determine clinical outcome, including pathologic complete response rate, post-treatment pathologic downstaging rate, recurrence-free survival (RFS), overall survival (OS) and neoadjuvant rectal score, among patients who are treated with standard neoadjuvant chemoradiation or TNT, with an aim to investigate how baseline biomarkers and changes in biomarkers with standard therapies may be associated with, and modulate, clinical outcomes.

DETAILED DESCRIPTION:
At enrollment, subjects should be planned to receive either neoadjuvant chemoradiation or total neoadjuvant therapy, with the choice of regimen at the discretion of treating investigators. Subjects will have been staged as deemed consistent with standard of care, including either a pelvic Magnetic resonance imaging (MRI) and/or an endorectal ultrasound, and deemed to have either T3-T4 primary tumor or node-positive tumor.

Neoadjuvant Chemoradiation Subjects will undergo endoscopic tumor biopsy within 6 weeks of the start of standard of care chemoradiation. Subjects will also have a baseline peripheral blood sample collected.

Subjects will receive neoadjuvant chemoradiation per standard of care. This is typically comprised of radiotherapy with concurrent capecitabine 825 mg/m2 by mouth (po) two times daily (bid) (typically rounded to the nearest 500 mg dose) or infusional 5-fluorouracil (5FU). However, dosing and administration are at the discretion of the treating medical and radiation oncologist.

An acceptable alternative approach is short-course radiation therapy per standard of care, which is typically comprised of radiotherapy, with surgery within 1 week of completion of therapy or delayed for 6-8 weeks. Selection of the optimal radiation therapy approach is at the discretion of the treating medical oncologist, radiation oncologist, and surgical oncologist. However, generally, short-course radiation therapy is not recommended for low-lying tumors less than 5 centimeters (cm) from the anal verge.

Occasionally patients with inadequate response after neoadjuvant chemoradiation may be recommended to proceed with subsequent consolidative chemotherapy with 5-Fluorouracil, leucovorin, and oxaliplatin (mFOLFOX6) or capecitabine and oxaliplatin (CAPOX) for 16-18 weeks before surgical resection. This treatment is at the discretion of the treating medical oncologist, radiation oncologist, and surgical oncologist. These subjects will be allowed to remain on study.

Surgery will occur approximately 4-8 weeks after chemoradiation or consolidative chemotherapy, depending on clinical factors (i.e. resectability, presence or absence of metastatic disease), although it may occur as soon as 1 week after completing short-course radiation therapy. The timing of surgical resection after completion of neoadjuvant therapy is at the discretion of the treating surgical oncologist. At the time of surgery, tumor samples and peripheral blood samples for correlative studies will be collected.

Subjects who do not receive preoperative mFOLFOX6 or CAPOX typically receive postoperative adjuvant chemotherapy with a fluoropyrimidine +/- oxaliplatin for an additional 16-18 weeks of therapy, if permitted based on recovery after surgical resection and post-surgical performance status. This treatment is at the discretion of the treating medical oncologist. Subjects will remain on study regardless of postoperative therapy administration or duration.

Total Neoadjuvant Therapy Subjects will undergo endoscopic tumor biopsy within 6 weeks of the start of standard of care treatment with chemotherapy. Subjects will also have a baseline peripheral blood sample collected.

Subjects who are intended to receive total neoadjuvant therapy will typically receive chemotherapy with mFOLFOX6 or CAPOX for 16-18 weeks, followed by chemoradiation. Dosing and administration are at the discretion of the primary medical and radiation oncologist. Alternative subsequent approaches such as short-course radiotherapy are also acceptable at the discretion of the treating medical and radiation oncologist.

Surgery will occur approximately 4-8 weeks after chemoradiation depending on clinical factors (i.e. resectability, presence or absence of metastatic disease), although it may occur as soon as 1 week after completing short-course radiation therapy. The timing of surgical resection after completion of neoadjuvant therapy is at the discretion of the treating surgical oncologist. At the time of surgery, tumor samples and peripheral blood samples for correlative studies will be collected.

Duration of Therapy

The duration of therapy should be defined per the subject's standard of care. Reasons to discontinue treatment may include:

* Disease progression
* Inter-current illness that prevents further administration of treatment
* Unacceptable adverse event(s)
* Pregnancy
* Subject decides to withdraw from study treatment, or
* General or specific changes in the subject's condition render the subject unacceptable for further treatment in the judgment of the investigator.
* Subject has completed the treatment regimen
* Subject is lost to follow up

Duration of Follow Up After surgery, subjects will be followed with routine surveillance at the discretion of treating investigators. Subjects will be followed for survival and disease status for at least 3 years after surgery or until death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained to participate in the study and HIPAA authorization for release of personal health information.
* Age ≥ 18 years at the time of consent.
* ECOG (Eastern Cooperative Oncology Group) Performance Status of 0-2 (See Appendix A. ECOG Performance Status Scale).
* Histological or cytological confirmation of rectal adenocarcinoma.
* Planned to receive treatment with neoadjuvant therapy, comprised of either 1) chemoradiation with concurrent fluoropyrimidine or short-course radiotherapy, or 2) total neoadjuvant therapy with fluoropyrimidine +oxaliplatin followed by chemoradiation or short-course radiotherapy. Rectal adenocarcinoma patients deemed candidates for neoadjuvant therapy include:

  1. Tumor staged as T3-4 or node-positive by pelvic MRI or endorectal ultrasound, or node-positive by CT scan; OR
  2. Tumor fixed to extra colonic structures as determined by digital rectal examination; OR
  3. Tumor < 5 cm from sphincter mechanism.
* Willing and able to undergo baseline rectal tumor biopsy, and willing and able to donate blood for research purposes.
* Females of childbearing potential must be willing to abstain from heterosexual activity or to use 2 forms of effective methods of contraception from the time of informed consent until 12 weeks after treatment discontinuation. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method or an intrauterine device that meets <1% failure rate for protection from pregnancy in the product label.
* Male subjects with female partners must have had a prior vasectomy or agree to use an adequate method of contraception (i.e., double barrier method: condom plus spermicidal agent) starting with the first dose of study therapy through 12 weeks after the last dose of study therapy.
* Subjects are willing and able to comply with study procedures based on the judgement of the investigator or protocol designee.

Exclusion Criteria:

* Patients with colon carcinomas that are too proximal to receive neoadjuvant therapy per routine clinical practice (i.e. with primary tumor proximal to or at the sigmoid colon).
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
* Has a known additional malignancy that is active and/or progressive and is requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, or other cancer for which the subject Is not currently receiving anti-cancer therapy such as chemotherapy, radiation therapy, targeted therapy, immunotherapy, or hormonal therapy.
* Patients who are not candidates at the discretion of their treating physicians to receive neoadjuvant chemoradiation or total neoadjuvant therapy (e.g. poor performance status, significant comorbidities, clinically significant organ dysfunction).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
complete pathologic response (pCR) rate | At time of surgery (1- 26 weeks after completion of standard of care neoadjuvant treatment)
  Anatomic stage for rectal cancer uses the American Joint Committee on Cancer (AJCC) Tumor/Node/Metastasis (TNM) system, which is based on:Size of primary tumor (T) and whether it has grown into nearby areas. Spread to regional lymph nodes (N). Spread (metastasis; M) to other organs of the body. Once the T, N, and M categories have been determined, this information is combined into a prognostic group. Higher numbers mean the cancer is more advanced. Stage prefixes include "c" for clinical stage, "p" for pathological stage, and "y" to indicate that the clinical or pathologic classification has been determined after preoperative therapy
  Complete pathologic response is defined as no disease on pathology at resection (ypT0N0).

SECONDARY OUTCOMES:
pathologic down staging rate | At time of surgery (1-26 weeks after completion of standard of care neoadjuvant treatment)
  Defined as a decrease in Tumor (T) and/or Nodal (N) stage from baseline to pathologic post-treatment determination, without any increase in T, N, or M stage.
near pathological complete response (near-pCR) rate | At time of surgery (1-26 weeks after completion of standard of care neoadjuvant treatment)
  Near-pCR will be defined as minimal tumor on pathology at resection (ypT0-1 N0).
R0 resection rate | At time of surgery (1-26 weeks after completion of standard of care neoadjuvant treatment)
  R0 resection will be defined as resection of all appreciable disease with a margin > 1 millimeter (mm) distally, proximally, and radially/circumferentially.
Recurrence Free Survival (RFS) rate | 3 years after surgical resection
  Defined as the time from day 1 of neoadjuvant chemotherapy until definitive local or metastatic disease recurrence or death as a result of any cause.
Overall Survival (OS) rate | 3 years after surgical resection
  Defined as the time from day 1 of neoadjuvant chemotherapy until death as a result of any cause.
Median Neoadjuvant Rectal Score (NAR) | At time of surgery (1-26 weeks after completion of standard of care neoadjuvant treatment)
  With clinical T stage (cT) comprised of 1, 2, 3, or 4; pathologic T stage (pT) comprised of 0, 1, 2, 3, or 4; and pathologic N stage (pN) comprised of 0, 1, or 2 (according to AJCC clinical rectal staging criteria)., the Neoadjuvant rectal score (NAR)will be calculated after resection as follows:
  NAR = [5 pN - 3 (cT-pT) + 12]2 / 9.61
  A higher score indicates poorer prognosis

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Lee, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials